CLINICAL TRIAL: NCT04743063
Title: Prospective Monitoring of Angiotensin Receptor Neprilysin Inhibitor in Older Adults With Heart Failure and Frailty
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Dae Hyun Kim, MD, MPH, ScD, Associate Professor, Brigham and Women's Hospital
Other Study IDs: 2019P000110-ARNI
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Heart Failure, Systolic; Frailty
MeSH Terms: conditions — Heart Failure, Systolic; Frailty | interventions — sacubitril and valsartan sodium hydrate drug combination; Angiotensin Receptor Antagonists; azilsartan; candesartan; eprosartan; Irbesartan; Losartan; olmesartan; Telmisartan; Valsartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- New users of angiotensin receptor neprilysin inhibitor
  Interventions: Drug: sacubitril/valsartan
- New users of angiotensin II receptor blockers
  Interventions: Drug: Angiotensin II Receptor Blockers

INTERVENTIONS:
Drug: sacubitril/valsartan — Initiation of sacubitril/valsartan, identified using prescription fill in pharmacy claims
  Groups: New users of angiotensin receptor neprilysin inhibitor
Drug: Angiotensin II Receptor Blockers — Initiation of ARBs, identified using prescription fill in pharmacy claims
  Other Names: azilsartan; candesartan; eprosartan; Irbesartan; losartan; Olmesartan; telmisartan; valsartan
  Groups: New users of angiotensin II receptor blockers

SUMMARY:
The objective of this study is to establish a near-real-time prospective monitoring program in Medicare, Optum and MarketScan Research data to evaluate the benefit of new cardiovascular disease (CVD) drugs for older adults with frailty. Prospective monitoring program seeks to find early effectiveness and safety signals of new drugs by updating the analysis at regular intervals as new Medicare data become available. This study specifically aims to emulate a prospective surveillance of the effectiveness and safety of Angiotensin Receptor Neprilysin Inhibitor(ARNI) vs. a comparator, Angiotensin II Receptor Blockers (ARBs), in older adults with Heart Failure with Reduced Ejection Fraction (HFrEF) and different frailty status. This program will be enhanced by incorporating a novel claims-based frailty index, which has been shown useful in assessing how the benefits and harms of drug therapy vary by frailty.

DETAILED DESCRIPTION:
Data sources of use for this study are: Medicare Database, Optum Database, and MarketScan Research Database. All data from years 2014-2020 will be included in the study.

This study follows a sequential cohort monitoring design. The monitoring analysis will include 1) retrospective analysis of available data (2015-2017) at the time of first analysis (January 2021) and 2) prospective analysis of new data (2018-2020) as they become available to the researchers. Within each database, we will emulate biannual updating of data by creating a propensity score (PS)-matched cohort of new users every 6-month interval, beginning on the first marketing of ARNI (July 7, 2015-December 31, 2015, and 6-month intervals afterwards). Each sequential cohort will be followed for development of the outcomes of interest. Outcome analysis will be performed at a pre-specified 6-month interval (prospective analysis). The surveillance will be performed by frailty status (frail vs non-frail) at the time of drug initiation. The results from each database will be pooled using fixed-effects meta-analysis (assuming low heterogeneity across the databases).

ELIGIBILITY:
Inclusion Criteria:

* Continuous enrollment for medical and drug insurance (e.g., Medicare Part A, B, and D) in [-365, 0] days
* Diagnosis of Heart Failure either two outpatient diagnosis or one inpatient diagnosis in [-365, 0] days
* Reduced Ejection Fraction < 45% identified using a validated claims-based algorithm in [-365, 0] days

  * Day 0 is the initiation date of the study drug.

Exclusion Criteria:

* No prior use of Angiotensin receptor neprilysin inhibitor or angiotensin II receptor blocker in [-365, -1] days
* No recent HF hospitalization, defined as HF diagnosis (defined in attached protocol) in the primary position in the inpatient dataset in [-60, 0] days
* No recent nursing facility stay (defined in attached protocol) for [-60, 0] days
* Age < 65 years
* Exposure to both drugs on day 0
* Contraindication to either drug (exclusion assessment window: [-60, 0] days, unless specified otherwise; algorithms specified in attached protocol)

Note: If a patient meets the above-mentioned eligibility criteria more than once, only the first record will be included.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Study population includes older patients with heart failure with reduced ejection fraction who initiates an angiotensin receptor neprilysin inhibitor or an angiotensin II receptor blocker.
Sampling Method: Non-Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with composite events of death or heart failure hospitalization | July 2015 - December 2020
  All-cause mortality OR heart failure hospitalization
Number of patients with composite serious adverse events | July 2015 - December 2020
  Hypotension OR acute kidney injury/acute kidney failure OR hyperkalemia OR angioedema

SECONDARY OUTCOMES:
Number of patients with all-cause mortality | July 2015 - December 2020
  All-cause mortality is defined by the National Death Index file or vital status information in the claims dataset.
Number of patients with heart failure hospitalization | July 2015 - December 2020
  Heart failure hospitalization is defined as any hospitalization with relevant diagnosis codes in the primary position.
Number of patients with hypotension | July 2015 - December 2020
  Hypotension is defined as any hospitalization or Emergency Department visit with relevant diagnosis codes in the primary position.
Number of patients with hyperkalemia | July 2015 - December 2020
  Hyperkalemia is defined as any hospitalization or Emergency Department visit with relevant diagnosis codes in the primary position.
Number of patients with acute kidney injury/acute kidney failure | July 2015 - December 2020
  Acute kidney injury/Acute kidney failure is defined as any hospitalization or Emergency Department visit with relevant diagnosis codes in the primary position.
Number of patients with angioedema | July 2015 - December 2020
  Angioedema is defined as any hospitalization or Emergency Department visit with relevant diagnosis codes in the primary position.

CONTACTS AND LOCATIONS:
Overall Officials: Dae Hyun Kim, MD, MPH, ScD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham And Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/63/NCT04743063/Prot_001.pdf